CLINICAL TRIAL: NCT03182322
Title: An Immune Efficacy Study for Primary Prevention Using Intranasal Insulin Therapy in Islet Autoantibody Negative Children at High Genetic Risk for Type 1 Diabetes
Brief Title: PINIT Study: Primary Intranasal Insulin Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Technische Universität Dresden (Other); Ludwig-Maximilians - University of Munich (Other); Helmholtz Zentrum München (Industry); University Hospital Carl Gustav Carus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 808040015
Record Dates: First submitted 2017-03-08; First posted 2017-06-09 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; T1D; diabetes mellitus; intranasal insulin; mucosal tolerance; autoantigen; self tolerance; prevention; at risk for developing type 1 diabetes; juvenile diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intranasal insulin (Experimental): rH-insulin formulation and for a dose of 440 IU insulin to the nasal mucosa. Treatment will be administered daily for the first 7 intervention days, and one day per week thereafter for 6 months.
  Interventions: Drug: intranasal insulin
- intranasal placebo (Placebo Comparator): Treatment with placebo nasal spray daily for the first 7 intervention days and one day per week thereafter for 6 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: intranasal insulin — Total of 6 months treatment; daily for the first 7 intervention days and one day per week thereafter (formulation containing rH-insulin, benzalkonium chloride, glycerol and water)
  Arms: intranasal insulin
Other: Placebo — Total of 6 months treatment; daily for the first 7 intervention days and one day per week thereafter placebo (formulation containing benzalkonium chloride, glycerol and water)
  Arms: intranasal placebo

SUMMARY:
Type 1 diabetes (T1D) results from an autoimmune destruction of the insulin-producing beta cells. Administration of mucosal insulin in islet autoantibody-negative children who are genetically predisposed for T1D offers the potential for inducing immunological tolerance to beta cells and thereby protect against the development of islet autoimmunity and T1D. Intranasal insulin has the advantage that whole protein will be exposed at the mucosa. Therefore, the available dose of insulin when administered intranasally is likely to be consistent between individuals. On this basis, the investigators aim to conduct a placebo-controlled, double-blind/double-masked primary intervention pilot trial (PINIT Study) of intranasal insulin treatment in islet autoantibody negative children to test immune efficacy and safety in the primary prevention setting. This pilot will help to develop and design a Phase III study aiming to test efficacy of preventing islet autoimmunity and T1D.

DETAILED DESCRIPTION:
Hypothesis: The hypothesis is that intranasal administration of insulin will induce protective immune responses and prevent T1D-autoimmunity, and the development of T1D.

Objectives: To determine whether intranasal administration of 440 IU insulin to children with high genetic risk for T1D will induce likely protective IgG or IgA antibody responses to insulin, and/or T-cell responses to insulin and/or proinsulin.

Intranasal insulin will be applied as a fine aerosol spray to the back of the nose. The insulin formulation and method of administration of intranasal insulin is designed to stimulate local mucosal immunity to insulin as an antigenic protein. Without an absorption enhancer, such as a surfactant, intranasal insulin is not anticipated to have systemic hormonal effects. The presentation is a multi-dose spray device with nasal actuator in a brown glass vial designed to deliver 50 μl spray doses to the nasal mucosa.

The PINIT Study is designed as a randomized, placebo-controlled, double-blind, multicenter, primary intervention pilot phase II study, in which intranasal insulin will be administered daily for the first seven days and once per week thereafter. The study will include 38 islet autoantibody negative children with the HLA DR3/4-DQ8 genotype or with a first degree relative with T1D and at least one HLA DR4-DQ8 haplotype and no protective HLA DR-DQ alleles or haplotypes. These 38 children will be randomized to either insulin or placebo in a 1:1 ratio. The study will be monitored by an external Data Safety Monitoring Committee (DSMB).

Recruitment will be carried out German wide and will be organized by clinical centers in Munich and Dresden. PINIT will determine the immune bioavailability of mucosal insulin to the immune system in the age group of 1 year to 7 years and assess safety of treatment with intranasal insulin at a single dose (440 IU).

Primary outcome - immune efficacy: The primary outcome is immune efficacy measured by the activation of an immune response (antibody or CD4+ T cell) against insulin.

Additional outcomes are:

* safety assessed by blood glucose concentrations in the first 2 hours after receiving study drug to determine whether the treatment induces hypoglycaemia, and the development of islet autoantibodies to GAD and IA-2 and ZnT8 is assessed at 3 and 6 months after commencing treatment.
* mechanistic T cell studies to determine the characteristics of any T cell response to insulin.
* Flow cytometry to measure T cell and monocyte subpopulations
* RNA seq on peripheral blood mononuclear cells
* Serum inflammatory markers

Comparisons between treatment groups will be performed on the whole cohort and also separately on the participants by the type 1 diabetes susceptible INS genotype, and after stratification for age and SIGLEC1 (CD169) positivity of monocytes.

Time schedule: The recruitment phase will run over a period of 12 months. Enrolled participants will be treated for 6 months. First patient first visit (FPFV) occured in May 2018 and the last patient last visit (LPLV) occured on 18. August 2020. The overall end of trial time point is defined as the time when all mechanistic assays and measurement of lab values including T-cell stimulation tests have been completed. This is expected by end of February 2021.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 1 year to 7 years (randomization must be performed prior to 8th birthday) who

   * have the HLA DR3-DQB1*0201/DR4-DQB1*0302 or the HLA DR3-DQB1*0201/DR4-DQB1*0304 genotype or
   * have a first degree relative with type 1 diabetes, and have a HLA genotype that includes the HLA DR4-DQB1*0302 or HLA DR4-DQB1*0304 haplotype, and does not include one of the following alleles DR 11, DR 12, DQB1*0602, or haplotypes DR7-DQB1*0303, DR14-DQB1*0503, DR13-DQB1*0603 and must be
2. Islet autoantibody negative (autoantibodies against insulin, GAD, IA-2 and ZnT8) at time of screening.

Exclusion Criteria:

1. Concomitant disease or treatment, which may interfere with assessment or cause immunosuppression, as judged by the investigators.
2. Any condition that could be associated with poor compliance.
3. Any defect or pathology of nasal passage, which would preclude application of the intranasal spray.
4. Any moderate to severe intolerance to ingredients of the investigational medicinal product.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
The activation of an immune response (antibody or CD4+ T cell) against insulin. | change from baseline (visit 1) in CD4+ T cell response measured as a stimulation index at 3 months (visit 2) and 6 months (visit 3) of treatment
  The responses are as previously defined in the Pre-POINT study (JAMA 313:1541-9). An antibody response is defined as serum IAA positivity in the competitive immuno-precipitation assay, an increase from baseline (>10 cpm) in serum IgG binding to insulin, or a positive salivary IgA binding to insulin. A CD4+ T cell response is defined as a stimulation index >3 and a >2-fold increase from stimulation index at baseline. A positive response (responder) will be defined as a child with an antibody or T cell response to insulin at any time point during treatment. The number of responders in the insulin treated group will be compared with the number of responders in the placebo treated group.

OTHER OUTCOMES:
Hypoglycemia | Measured at baseline (visit 1) and at each subsequent visit at 3 months (visit 2) and 6 months (visit 3) of treatment.
  Metabolic changes within two hours after receiving study drug. This will be performed at the first administration of intranasal insulin or placebo at baseline, 3 months and 6 months of treatment (visit 1, visit 2, and visit 3). At these visits, blood glucose concentrations will be measured at 0 minutes, 30 minutes, 60 minutes, and 120 minutes after receiving study drug to determine whether the treatment induces hypoglycaemia which is defined as <50 mg/dl.
GAD, IA-2 and ZnT8 autoantibodies | Measured at baseline and at 3 months, 6 months.
  The purpose is to detect seroconversion to islet autoantibody positive. Measurements are performed using a radiobinding immunoprecipitation assay. Frequency of confirmed positive autoantibody results (i.e. autoantibody positive in two consecutive serum samples) will be compared between placebo vs. insulin treated children
Gene expression analysis of single cells. | baseline, 3 months and 6 months
  The gene expression of the insulin responsive cells will be compared between the placebo and study drug treated children using different multivariable gene expression analysis methods (for instance Stochastic Neighbor Embedding (tSNE) analysis).
FOXP3/IFNG signature ratio | baseline, 3 months and 6 months
  The FOXP3 signature/IFNG signature ratio of the insulin responsive cells will be compared between the placebo and study drug treated children.
Change in IgG-IAA | baseline, 3 months and 6 months
  The change from baseline in IgG-IAA measured by radio-binding assay will be compared between placebo and study drug treated children.
Antibody responses | baseline,3 months and 6 months
  Antibody responses will be compared between placebo and study drug treated children using time to event analyses.
CD4+ T cells responses to insulin | baseline, 3 months and 6 months
  CD4+ T cells responses to insulin will be compared between placebo and study drug treated children using time to event analyses.
CD4+ T cells responses to pre-proinsulin peptides | change from baseline to 3 months and 6 months
  CD4+ T cells responses to pre-proinsulin peptides will be compared between placebo and study drug treated children using time to event analyses.
CD8+ T cell responses to insulin | baseline, 3 months and 6 months
  CD8+ T cell responses to insulin using the definition for CD4+ T cells as defined above will be compared between placebo and study drug treated children using time to event analyses.
CD8+ T cells responses to pre-proinsulin peptides | baseline, 3 months and 6 months
  CD8+ T cells responses to pre-proinsulin peptides will be compared between placebo and study drug treated children using time to event analyses.
T cell and monocyte populations | baseline, 3 months and 6 months
  Peripheral blood T cell and monocyte populations will be compared between placebo and study drug treated children.
Plasma inflammatory markers | baseline, 3 months and 6 months
  Plasma inflammatory markers will be compared between placebo and study drug treated children.Therefore, the Olink Target 96 Inflammation protein biomarker panel is used. An overview of all 92 biomarkers can be seen on the following homepage: https://www.olink.com/products/inflammation/
Transcriptome of peripheral blood cell populations | baseline, 3 months and 6 months
  If available, transcriptome of peripheral blood cell populations will be compared between placebo and study drug treated children.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Achenbach, PD Dr., Principal Investigator — Forschergruppe Diabetes, Klinikum rechts der Isar, Technische Universität München, Lehrstuhl für Diabetes und Gestationsdiabetes, der Technischen Universität München, Kölner Platz 1, 80804 München, Germany; Anette-G. Ziegler, Prof. Dr., Principal Investigator — Forschergruppe Diabetes, Klinikum rechts der Isar, Technische Universität München, Lehrstuhl für Diabetes und Gestationsdiabetes, der Technischen Universität München, Kölner Platz 1, 80804 München, Germany
Locations (2):
- Germany (2):
  - Klinik und Poliklinik für Kinder und Jugendmedizin, Universitätsklinikum Carl Gustav Carus, Technische Universität Dresden, Fetscherstraße 74, 01307 Dresden, Germany, Dresden
  - Forschergruppe Diabetes, Klinikum rechts der Isar, Technische Universität München, Lehrstuhl für Diabetes und Gestationsdiabetes der Technischen Universität München, München

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.helmholtz-muenchen.de/idf1